CLINICAL TRIAL: NCT02347202
Title: Tools for Distance Delivery of an Evidence-based AD Family Caregiver Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-01185
Record Dates: First submitted 2015-01-09; First posted 2015-01-27 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Counseling
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Health Services Needs and Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online counseling via Zoom teleconferencing (Experimental): Each participant will be assigned a random number which is linked to group assignment. The numbers will be assigned consecutively to participants as they enroll. All caregivers in the treatment group will receive 6 counseling sessions in 4 months, using teleconferencing. The first session will be an individual session. The caregiver will be asked to select family members to participate in the next 4 sessions. The 4 family sessions will be followed by another individual session with the spouse/partner caregiver. The counselor will send the primary caregiver an email to be forwarded to family members with instructions on how to access the TTDC training on using the teleconferencing technology. All caregivers in the control group will be able to call the counselor for resource information and support.
  Interventions: Other: Online counseling via Zoom teleconferencing
- Telephone support as needed (Other): All caregivers in the control group will be able to call the counselor for resource information and support as needed.
  Interventions: Other: Telephone support as needed

INTERVENTIONS:
Other: Online counseling via Zoom teleconferencing
  Arms: Online counseling via Zoom teleconferencing
Other: Telephone support as needed
  Arms: Telephone support as needed

SUMMARY:
A 20+ year randomized controlled trial (RCT) demonstrated the many benefits of a counseling and support intervention for spouse caregivers, the NYU Caregiver Intervention (NYUCI). The NYU Caregiver Intervention (NYUCI) is an evidence-based intervention that provides counseling and support for families involved in the care of a relative or friend with Alzheimer's Disease and Related Dementias (ADRD). Most notably, the NYUCI substantially reduced caregiver's depressive symptoms, improved their physical health, and extended the time persons with ADRD remained at home by an average of 1.5 years (Mittelman et al., AG14634, formerly MH42216; See http://www.ncbi.nlm.nih.gov/pubmed/17101889).

The intervention is now being widely implemented in-person, but there are barriers that prevent many caregivers from receiving its benefits, including geographic distance; impediments to older adults leaving their homes; and travel considerations for counselors which make it impossible to provide the NYUCI in person.

The goal of this study is to evaluate the efficacy of an online videoconferencing version of the NYUCI. This innovative application has massive implications for social service delivery to older adults, because it will make it possible to deliver an in-person intervention, via the internet, which is already evidenced based to older adult caregivers who cannot currently be served. It will create the online reservation and management technology linking counselors with families as well as the evidence of effectiveness of providing such services via secure video teleconferencing vehicles. The proposed Telehealth Technology for Distance Counseling (TTDC) and related online educational training modules will connect skilled providers to the families of persons with dementia without regard to geographic location. Implications for rural healthcare delivery are particularly persuasive. To the investigators knowledge, this will be the first large-scale TTDC to be developed and rigorously tested with a randomized controlled trial. The investigators hypothesize that such a system, coupled with online training for providers and families on tele- counseling and distance caregiving, will have similar benefits to those achieved with in-person counseling during the original NYUCI RCT.

This project includes an online reservation and management technology linking counselors with families via secure videoconferencing vehicles. The Telehealth Technology for Distance Counseling (TTDC), and online technology developed as part of this overall effort, will connect skilled providers to the families of persons with dementia without regard to geographic location. The related online clinical modules (i.e., interactive, computer-based educational materials) developed as a part of this grant effort will prepare counselors to provide the intervention, and caregivers to utilize the internet software, to be able to participate in counseling.

The TTDC will include a scheduling system to link counselors to families at their mutual convenience and assure delivery in a cost-effective manner. The TTDC has the additional potential to transform ADRD care in ethnic and culturally diverse communities by connecting highly trained NYUCI counselors with specialized language and cultural skills to families who would not have access to these resources locally.

In this study investigators will have 240 caregivers navigate the online educational module and the online reservation system for connecting caregivers with social workers. Half of the caregivers will then be paired with social service providers to receive counseling over the telephone, and the other half with be paired with social service providers to receive counseling via Zoom, a video conferencing program. Recruiting across the United States and Toronto, Canada.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for caregivers to become research participants include:

1. access to an Internet-connected computer with a camera, microphone, and speakers either at home, or at another location that affords privacy;
2. fluent in spoken and written English; and
3. caregivers who participate must be spouses or partners of people with dementia living with them at home when they enter the study. In addition, all caregivers must have at least one family member (or close friend) with whom they are in communication about the person with dementia, and/or their issues related to being a caregiver, who can participate in family counseling sessions; if not, they are excluded from the study.

Inclusion criteria for counselors to be research participants in both the pilot study and the RCT:

1. Certified or Master's level social worker, a nurse with an RN and at least two years' experience working with older adults and their family members evaluated on an individual basis by the PIs);
2. counselors who have received training online or in person in conducting the NYUCI and provided the intervention to at least one caregiver in person;
3. counselors who have completed the online training to conduct the NYUCI via videoconferencing;
4. counselors who have demonstrated the ability to contact caregivers and families via videoconferencing by interacting with HealthCare Interactive (HCI) staff in mock sessions (HCI is the technology developer for this Phase II effort); and
5. counselors who have confirmed they have personal liability and malpractice insurance.

Exclusion Criteria:

Exclusion criteria for caregivers to be participants are:

1. no access or severely limited access to an Internet-connected computer with a camera;
2. not fluent in spoken and written English;
3. not having a family member with whom they are in communication about the person with dementia; and
4. apparent severe mental or physical illness (e.g., self report of clinical depression).

Exclusion criteria for counselors include:

1. not a certified or Master's level social worker or nurse with an RN and at least two years' experience working with older adults and their family members, or other professional with at last two years' experience working with older adults and their family members (to be decided by the PIs);
2. counselors who have not received training online or in person in conducting the NYUCI;
3. counselors who have not completed the online training to conduct the NYUCI via videoconferencing;
4. counselors who cannot demonstrate ability to contact caregivers and families via videoconferencing by interacting with HCI; and
5. counselors who do not have personal liability and malpractice insurance.

Ages: 21 Years to 125 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Differences in depressive symptoms between groups (One-way analysis of variance, questionnaire) | Four, eight, and twelve months after intervention
  One-way analysis of variance to evaluate differences in depressive symptoms between groups. This data will be collected via a questionnaire.
Differences in reactions to problem behaviors between groups (questionnaire) | Four, eight, and twelve months after intervention
  This information will be collected via a questionnaire.
Differences in satisfaction with social support between groups (questionnaire) | Four, eight, and twelve months after intervention
  This information will be collected via a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Mittelman, DrPH, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- See also: Improving caregiver well-being delays nursing home placement of patients with Alzheimer disease. — http://www.ncbi.nlm.nih.gov/pubmed/17101889